CLINICAL TRIAL: NCT00088478
Title: A Double-Blind, Randomized Study Comparing Intramuscular Olanzapine Depot With Placebo in the Treatment of Patients With Schizophrenia
Brief Title: Comparison of Intramuscular Olanzapine Depot With Placebo in the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5984; F1D-MC-HGJZ
Record Dates: First submitted 2004-07-26; First posted 2004-07-28 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Intramuscular Olanzapine Depot
Drug: Placebo

SUMMARY:
Key objectives of this clinical study are to:

* Determine how well intramuscular (IM) olanzapine depot works compared to placebo
* Evaluate the safety and tolerability of IM olanzapine depot compared to placebo
* Evaluate different doses of IM olanzapine depot compared to placebo to identify the best dose(s).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have schizophrenia and be experiencing a psychotic episode
* Each patient must have a level of understanding sufficient to complete all tests and examinations required by the protocol, and to provide informed consent
* Patient must not have participated in a clinical trial of another investigational drug, including olanzapine, within 1 month (30 days) prior to the study entry
* Female patients must not be pregnant or breast-feeding
* Female patients must not be experiencing acute, serious or unstable medical conditions other than schizophrenia

Exclusion Criteria:

* Patients who were previously treated with olanzapine and are considered to be treatment-resistant to olanzapine, in the opinion of the investigator
* One or more seizures without a clear and resolved etiology is exclusionary. However, if the patient has had one or more seizures in the past with an identifiable etiology, and that etiology has been resolved, the patient may be entered.
* Treatment with clozapine within 4 weeks prior to visit 1
* DSM-IV or DSM-IV-TR substance (except nicotine and caffeine) dependence within the past 30 days
* Treatment with remoxipride within 6 months (180 days) prior to visit 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2004-06; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Demonstrate superiority of IM olanzapine depot 300 mg/2 weeks, 405 mg/4 weeks, and 210 mg/2 weeks dosages compared with placebo in the treatment of patients with schizophrenia

SECONDARY OUTCOMES:
To assess the efficacy of 300 mg/2 weeks, 405 mg/4 weeks, and 210 mg/2 weeks IM olanzapine depot compared with placebo in CGI-I
To determine the earliest time point at which 300 mg/2 weeks, 405 mg/4 weeks, and 210 mg/2 weeks IM olanzapine depot show superior clinical improvement compared with placebo
To assess the efficacy of 300 mg/2 weeks, 405 mg/4 weeks, and 210 mg/2 weeks IM olanzapine depot compared with placebo in CGI-S
To assess the efficacy of 300 mg/2 weeks, 405 mg/4 weeks, and 210 mg/2 weeks IM olanzapine depot compared with placebo in terms of change in PANSS Positive, PANSS Negative and PANSS General Psychopathology subscales
To assess the efficacy of 300 mg/2 weeks, 405 mg/4 weeks, and 210 mg/2 weeks IM olanzapine depot compared with placebo in change from baseline to endpoint in quality of life
To evaluate the safety and tolerability of 300 mg/2 weeks, 405 mg/4 weeks, and 210 mg/2 weeks IM olanzapine depot compared with placebo
To characterize the pharmacokinetics of olanzapine following multiple dosing with IM olanzapine depot at each of the prescribed dosing regimens

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (34):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Rosemead, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Santa Ana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Saint Louis, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Lawrence, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Chagrin Falls, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Norristown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Travelers Rest, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Kirkland, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Kirkland, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Zagreb, Croatia
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Saint Petersburg

REFERENCES:
- [Derived] Atkins S, Detke HC, McDonnell DP, Case MG, Wang S. A pooled analysis of injection site-related adverse events in patients with schizophrenia treated with olanzapine long-acting injection. BMC Psychiatry. 2014 Jan 14;14:7. doi: 10.1186/1471-244X-14-7. PMID 24423017
- [Derived] Detke HC, Zhao F, Witte MM. Efficacy of olanzapine long-acting injection in patients with acutely exacerbated schizophrenia: an insight from effect size comparison with historical oral data. BMC Psychiatry. 2012 May 30;12:51. doi: 10.1186/1471-244X-12-51. PMID 22646847
- [Derived] Witte MM, Case MG, Schuh KJ, Ascher-Svanum H. Effects of olanzapine long-acting injection on levels of functioning among acutely ill patients with schizophrenia. Curr Med Res Opin. 2012 Mar;28(3):315-23. doi: 10.1185/03007995.2012.657300. Epub 2012 Jan 31. PMID 22236137
- [Derived] Ascher-Svanum H, Zhao F, Detke HC, Nyhuis AW, Lawson AH, Stauffer VL, Montgomery W, Witte MM, McDonnell DP. Early response predicts subsequent response to olanzapine long-acting injection in a randomized, double-blind clinical trial of treatment for schizophrenia. BMC Psychiatry. 2011 Sep 23;11:152. doi: 10.1186/1471-244X-11-152. PMID 21943257
- [Derived] McDonnell DP, Detke HC, Bergstrom RF, Kothare P, Johnson J, Stickelmeyer M, Sanchez-Felix MV, Sorsaburu S, Mitchell MI. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, II: investigations of mechanism. BMC Psychiatry. 2010 Jun 10;10:45. doi: 10.1186/1471-244X-10-45. PMID 20537130
- [Derived] Detke HC, McDonnell DP, Brunner E, Zhao F, Sorsaburu S, Stefaniak VJ, Corya SA. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, I: analysis of cases. BMC Psychiatry. 2010 Jun 10;10:43. doi: 10.1186/1471-244X-10-43. PMID 20537128
- [Derived] Lauriello J, Lambert T, Andersen S, Lin D, Taylor CC, McDonnell D. An 8-week, double-blind, randomized, placebo-controlled study of olanzapine long-acting injection in acutely ill patients with schizophrenia. J Clin Psychiatry. 2008 May;69(5):790-9. doi: 10.4088/jcp.v69n0512. PMID 18452346
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com